CLINICAL TRIAL: NCT03202017
Title: A Pilot Study of Lung Volume Recruitment Combined With Expiratory Muscle Strength Training in ALS
Brief Title: Lung Volume Recruitment Combined With Expiratory Muscle Strength Training in ALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NEUR-2017-25778
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expiratory Muscle Strength Testing (EMST) (Active Comparator): EMST is a treatment method that has been used to improve cough function and swallowing in ALS. EMST uses a training device that has a valve set to 50% of a patient's maximum expiratory pressure (MEP). The patient exhales forcefully until the valve releases. Patients perform 5 sets of 5 repetitions a day, 5 days a week.
  Interventions: Procedure: Expiratory Muscle Strength Training (EMST)
- EMST + Lung Volume Recruitment (LVR) (Active Comparator): EMST is a treatment method that has been used to improve cough function and swallowing in ALS. EMST uses a training device that has a valve set to 50% of a patient's maximum expiratory pressure (MEP). The patient exhales forcefully until the valve releases. Patients perform 5 sets of 5 repetitions a day, 5 days a week.
  LVR is a technique to increase cough function that is performed with a resuscitation bag fitted with a mouthpiece and a one-way valve. The bag is used to expand the lungs, after which the patient makes a voluntary cough.
  Interventions: Procedure: EMST + Lung Volume Recruitment (LVR)

INTERVENTIONS:
Procedure: Expiratory Muscle Strength Training (EMST) — EMST uses a training device that has a valve set to 50% of a patient's maximum expiratory pressure (MEP). The patient exhales forcefully until the valve releases. Patients perform 5 sets of 5 repetitions a day, 5 days a week.
  Arms: Expiratory Muscle Strength Testing (EMST)
Procedure: EMST + Lung Volume Recruitment (LVR) — EMST uses a training device that has a valve set to 50% of a patient's maximum expiratory pressure (MEP). The patient exhales forcefully until the valve releases. Patients perform 5 sets of 5 repetitions a day, 5 days a week.
  LVR is a technique to increase cough function that is performed with a resuscitation bag fitted with a mouthpiece and a one-way valve. The bag is used to expand the lungs, after which the patient makes a voluntary cough. Half of the participants will perform the LVR technique in addition to the ESMT technique.
  Arms: EMST + Lung Volume Recruitment (LVR)

SUMMARY:
The purpose of this study is to investigate the effects of two treatment techniques called Expiratory Muscle Strength Training (EMST) and Lung Volume Recruitment (LVR) on breathing, swallowing, speech, and cough function in persons with mild to moderate ALS. Half of the participants will do EMST alone, and the other half of the participants will do EMST and LVR.

ELIGIBILITY:
Inclusion Criteria:

* ALS defined as possible, laboratory-supported probable, probable, or definite by El Escorial criteria
* Reduced Maximal Expiratory Pressure (MEP) compared to norms for age and sex
* Forced Vital Capacity (FVC) > 65% predicted

Exclusion Criteria:

* Inability to provide informed consent
* Relative contraindications to LVR, including known pneumothorax, active internal bleeding, unstable hypertension, unstable angina, emphysema, recent barotrauma, or FEV1 (Forced Expiratory Volume, trial 1)/FVC ratio < 0.7.
* Use of EMST or breath stacking > 3 days/week within 12 weeks of screening
* Amyotrophic Lateral Sclerosis-Cognitive Behavioral Scale (ALS-CBS) score predictive of dementia (≤ 10)
* Participation in another clinical trial of an intervention in ALS within 30 days of study enrollment or during study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Peak Cough Flow | Baseline (Week 0), Week 6, and Week 12
  Ventilatory measure that assesses the change in coughing ability at Baseline (Week 0), Randomization (Week 6), and End of Study (Week 12)

SECONDARY OUTCOMES:
Maximal Expiratory Pressure | Week 0, Week 6, Week 8, Week 10, and Week 12
  Measurement of respiratory muscle strength changes at Baseline (Week 0), Randomization (Week 6), Week 8, Week 10, and End of Study (Week 12)
Forced Vital Capacity | Baseline (Week 0), Week 6, and Week 12
  Measurement of changes in how much air is exhaled over a series of forced breaths at Baseline (Week 0), Randomization (Week 6), and End of Study (Week 12)
Eating Assessment Tool - 10 (EAT-10) | Baseline (Week 0), Week 6, and Week 12
  10-item patient reported outcome assessing changes in swallowing function at Baseline (Week 0), Randomization (Week 6), and End of Study (Week 12)
Swallowing Related Quality of Life (SWAL-QOL) | Baseline (Week 0), Randomization (Week 6), and End of Study (Week 12)
  44-item patient reported outcome assessing changes in swallowing impairment at Baseline (Week 0), Randomization (Week 6), and End of Study (Week 12)
Speech Intelligibility Test (SIT) | Baseline (Week 0), Randomization (Week 6), and End of Study (Week 12)
  Standardized assessment of speech intelligibility and efficiency in neuromuscular disorders. Measures changes in speech intelligibility at Baseline (Week 0), Randomization (Week 6), and End of Study (Week 12).

CONTACTS AND LOCATIONS:
Overall Officials: David Walk, MD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No